CLINICAL TRIAL: NCT07131735
Title: Intraoperative Detection of Breast Cancer by Electrosurgical Gas Analysis and Artificial Intelligence
Status: Recruiting | Type: Observational
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Sponsor
Other Study IDs: 230719001
Record Dates: First submitted 2025-07-28; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; odors and cancer; breast surgery; intraoperative margin assistant; artificial intelligence
MeSH Terms: conditions — Breast Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who have undergone conservative breast cancer surgery: This group will undergo an analysis of gases emitted by cauterization. This intervention will not modify the duration of the surgery, nor will it alter the patient's treatment and prognosis. The gases will be analyzed through the detection device, which will not have direct contact with the patient and will not influence the surgical outcomes of the resection surgery. The patient will be followed for 2 years through their clinical care records in the UC Christus health network, looking for the occurrence of disease recurrence.

SUMMARY:
The aim of this clinical trial is to assess the feasibility of training a device capable of distinguishing various gases emitted by tissues cauterized by an electrosurgical unit during a breast cancer resection surgery. The patients to be enrolled will be women over 18 years old diagnosed with breast cancer who are indicated for conservative breast cancer resection surgery as treatment.

The main questions to be answered are:

The specificity and sensitivity of the device in detecting margins compromised with tumor cells in resection surgeries.

Evaluate the applicability of the device in breast cancer surgeries for real-time detection of margins.

Evaluate the differences in the pattern of gases emitted in tumor cells vs normal cells.

By consenting, the study patients will allow the investigative team to access the clinical record, results of images, post-surgical biopsies, recording of the surgery while preserving the patient's anonymity, and the installation of the gas detection device. This device does not alter the flow of the surgery and does not add additional risk to it.

DETAILED DESCRIPTION:
The study will consist of measuring gases emitted during surgery. Prior to this, the device will be trained in the detection and recognition of the most prevalent gases in cancerous tissue. This will enable the AI to detect and classify cancerous breast tissue from healthy tissue. The study will include patients with different types and subtypes of breast cancer, such as ductal carcinoma in situ invasive ductal carcinoma, invasive lobular carcinoma, triple-negative breast cancer, human epidermal growth factor receptor 2 positive breast cancer, and hormone receptor-positive breast cancer. These types and subtypes reflect the diversity and complexity of breast cancer and may influence the performance and accuracy of the BCGC device.

During the clinical testing phase, the laboratory-acquired tissue detection capability will be evaluated in a real situation. For this, the device will be connected to a sterile PVC hose directly connected to a smoke extractor associated with the electrosurgical unit that will cauterize the tissues. To evaluate the sensitivity, specificity, and accuracy of the device, the AI's detection will be compared with the quick biopsy and the deferred biopsy of the surgical piece. For this, access will be obtained to the histological reports and the surgery will be recorded to identify margins.

The device will be calibrated once a month with gases of known nature, a maximum variability of 5% will be tolerated. If a greater variability is detected at the time of calibration, it will be changed to every 2 weeks. The information will be anonymized and stored on an SSD unit and will be deleted 5 years after the completion of the study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of malignant breast cancer
* Scheduled for BCS at the Hospital UC
* Able and willing to provide informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Patients with known hypersensitivity or allergy to any component of the BCGC device
* Participation in another interventional clinical trial within 30 days prior to enrolment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will recruit women from all over Chile who are indicated for conservative breast cancer surgery. It is estimated that the majority of patients will be those from Santiago de Chile who receive care from professionals in the UC Christus Health Network and decide to have surgery at the UC CHRISTUS Clinical Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-09-18 (Estimated); Study Completion 2025-09-18 (Estimated)

PRIMARY OUTCOMES:
Differentiation of cancerous tissue from normal tissue | Evaluation will be conducted 2 months post-surgery, comparing the biopsy results with the classification made by the device.
  Specificity, sensitivity, and accuracy of the device and software in tissue classification

SECONDARY OUTCOMES:
Applicability to the surgical workflow | The survey will be done 30 minutes after the conclusion of surgery and is estimated to require two minutes to complete.
  Installation time and the surgeon's subjective assessment will be measured using the "Device Applicability to Surgical Workflow" survey, which comprises three questions for a total score of 3-15 points. The survey will be administered once to each surgeon.
Biocompatibility | Adverse reactions will be evaluated from the moment of intervention up to 48 hours after the surgical procedure
  Biocompatibility of the materials used will be assessed by documenting adverse reactions during the surgical procedure and the immediate postoperative period.
Detecting volatile organic compounds in breast cancer tissue. | Measurement will occur intraoperatively from the surgeon's first electrosurgical incision until removal of the primary specimen-typically within the first hour of surgery. This timeframe applies to every analyzed procedure.
  The device is capable of real-time detection of organic compounds, with a latency not exceeding 1.5 seconds, and exhibits variable response slopes depending on the specific volatile organic compounds to which it is exposed.
Complications associated with the use of the device | Complications associated with device use will be assessed during the late postoperative period, defined as 48 hours after surgery up to one month post-intervention.
  Late complications related to device use will be assessed through reported occurrences.

CONTACTS AND LOCATIONS:
Locations (2):
- Chile (2):
  - Hospital Clínico UC CHRISTUS, Santiago, Santiago Centro
  - Facultad de medicina UC, Santiago, Santiago Metropolitan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McKinney SM, Sieniek M, Godbole V, Godwin J, Antropova N, Ashrafian H, Back T, Chesus M, Corrado GS, Darzi A, Etemadi M, Garcia-Vicente F, Gilbert FJ, Halling-Brown M, Hassabis D, Jansen S, Karthikesalingam A, Kelly CJ, King D, Ledsam JR, Melnick D, Mostofi H, Peng L, Reicher JJ, Romera-Paredes B, Sidebottom R, Suleyman M, Tse D, Young KC, De Fauw J, Shetty S. International evaluation of an AI system for breast cancer screening. Nature. 2020 Jan;577(7788):89-94. doi: 10.1038/s41586-019-1799-6. Epub 2020 Jan 1. PMID 31894144
- [Background] LeCun Y, Bengio Y, Hinton G. Deep learning. Nature. 2015 May 28;521(7553):436-44. doi: 10.1038/nature14539. PMID 26017442
- [Background] Keelan S, Flanagan M, Hill ADK. Evolving Trends in Surgical Management of Breast Cancer: An Analysis of 30 Years of Practice Changing Papers. Front Oncol. 2021 Aug 4;11:622621. doi: 10.3389/fonc.2021.622621. eCollection 2021. PMID 34422626
- [Background] Singla N, Dubey K, Srivastava V. Automated assessment of breast cancer margin in optical coherence tomography images via pretrained convolutional neural network. J Biophotonics. 2019 Mar;12(3):e201800255. doi: 10.1002/jbio.201800255. Epub 2018 Nov 13. PMID 30318761
- [Background] Ehteshami Bejnordi B, Veta M, Johannes van Diest P, van Ginneken B, Karssemeijer N, Litjens G, van der Laak JAWM; the CAMELYON16 Consortium; Hermsen M, Manson QF, Balkenhol M, Geessink O, Stathonikos N, van Dijk MC, Bult P, Beca F, Beck AH, Wang D, Khosla A, Gargeya R, Irshad H, Zhong A, Dou Q, Li Q, Chen H, Lin HJ, Heng PA, Hass C, Bruni E, Wong Q, Halici U, Oner MU, Cetin-Atalay R, Berseth M, Khvatkov V, Vylegzhanin A, Kraus O, Shaban M, Rajpoot N, Awan R, Sirinukunwattana K, Qaiser T, Tsang YW, Tellez D, Annuscheit J, Hufnagl P, Valkonen M, Kartasalo K, Latonen L, Ruusuvuori P, Liimatainen K, Albarqouni S, Mungal B, George A, Demirci S, Navab N, Watanabe S, Seno S, Takenaka Y, Matsuda H, Ahmady Phoulady H, Kovalev V, Kalinovsky A, Liauchuk V, Bueno G, Fernandez-Carrobles MM, Serrano I, Deniz O, Racoceanu D, Venancio R. Diagnostic Assessment of Deep Learning Algorithms for Detection of Lymph Node Metastases in Women With Breast Cancer. JAMA. 2017 Dec 12;318(22):2199-2210. doi: 10.1001/jama.2017.14585. PMID 29234806
- [Background] Chagpar AB, Killelea BK, Tsangaris TN, Butler M, Stavris K, Li F, Yao X, Bossuyt V, Harigopal M, Lannin DR, Pusztai L, Horowitz NR. A Randomized, Controlled Trial of Cavity Shave Margins in Breast Cancer. N Engl J Med. 2015 Aug 6;373(6):503-10. doi: 10.1056/NEJMoa1504473. Epub 2015 May 30. PMID 26028131
- [Background] Boppart SA, Luo W, Marks DL, Singletary KW. Optical coherence tomography: feasibility for basic research and image-guided surgery of breast cancer. Breast Cancer Res Treat. 2004 Mar;84(2):85-97. doi: 10.1023/B:BREA.0000018401.13609.54. PMID 14999139
- [Background] Assayag O, Antoine M, Sigal-Zafrani B, Riben M, Harms F, Burcheri A, Grieve K, Dalimier E, Le Conte de Poly B, Boccara C. Large field, high resolution full-field optical coherence tomography: a pre-clinical study of human breast tissue and cancer assessment. Technol Cancer Res Treat. 2014 Oct;13(5):455-68. doi: 10.7785/tcrtexpress.2013.600254. Epub 2013 Aug 31. PMID 24000981
- [Background] Tang R, Saksena M, Coopey SB, Fernandez L, Buckley JM, Lei L, Aftreth O, Koerner F, Michaelson J, Rafferty E, Brachtel E, Smith BL. Intraoperative micro-computed tomography (micro-CT): a novel method for determination of primary tumour dimensions in breast cancer specimens. Br J Radiol. 2016;89(1058):20150581. doi: 10.1259/bjr.20150581. Epub 2015 Nov 16. PMID 26568439
- [Background] Qiu SQ, Dorrius MD, de Jongh SJ, Jansen L, de Vries J, Schroder CP, Zhang GJ, de Vries EGE, van der Vegt B, van Dam GM. Micro-computed tomography (micro-CT) for intraoperative surgical margin assessment of breast cancer: A feasibility study in breast conserving surgery. Eur J Surg Oncol. 2018 Nov;44(11):1708-1713. doi: 10.1016/j.ejso.2018.06.022. Epub 2018 Jul 3. PMID 30005963
- [Background] McClatchy DM 3rd, Zuurbier RA, Wells WA, Paulsen KD, Pogue BW. Micro-computed tomography enables rapid surgical margin assessment during breast conserving surgery (BCS): correlation of whole BCS micro-CT readings to final histopathology. Breast Cancer Res Treat. 2018 Dec;172(3):587-595. doi: 10.1007/s10549-018-4951-3. Epub 2018 Sep 17. PMID 30225621
- [Background] Janssen NNY, van Seijen M, Loo CE, Vrancken Peeters MTFD, Hankel T, Sonke JJ, Nijkamp J. Feasibility of Micro-Computed Tomography Imaging for Direct Assessment of Surgical Resection Margins During Breast-Conserving Surgery. J Surg Res. 2019 Sep;241:160-169. doi: 10.1016/j.jss.2019.03.029. Epub 2019 Apr 23. PMID 31026794
- [Background] DiCorpo D, Tiwari A, Tang R, Griffin M, Aftreth O, Bautista P, Hughes K, Gershenfeld N, Michaelson J. The role of Micro-CT in imaging breast cancer specimens. Breast Cancer Res Treat. 2020 Apr;180(2):343-357. doi: 10.1007/s10549-020-05547-z. Epub 2020 Feb 4. PMID 32020431
- [Background] van Riet PA, Giorgio Arcidiacono P, Petrone M, Quoc Nguyen N, Kitano M, Chang K, Larghi A, Iglesias-Garcia J, Giovannini M, van der Merwe S, Santo E, Baldaque-Silva F, Bucobo JC, Bruno MJ, Aslanian HR, Cahen DL, Farrell J. Combined versus single use 20 G fine-needle biopsy and 25 G fine-needle aspiration for endoscopic ultrasound-guided tissue sampling of solid gastrointestinal lesions. Endoscopy. 2020 Jan;52(1):37-44. doi: 10.1055/a-0966-8755. Epub 2019 Jul 22. PMID 31330556
- [Background] Lange M, Reimer T, Hartmann S, Glass A, Stachs A. The role of specimen radiography in breast-conserving therapy of ductal carcinoma in situ. Breast. 2016 Apr;26:73-9. doi: 10.1016/j.breast.2015.12.014. Epub 2016 Feb 1. PMID 27017245
- [Background] Versteegden DPA, Keizer LGG, Schlooz-Vries MS, Duijm LEM, Wauters CAP, Strobbe LJA. Performance characteristics of specimen radiography for margin assessment for ductal carcinoma in situ: a systematic review. Breast Cancer Res Treat. 2017 Dec;166(3):669-679. doi: 10.1007/s10549-017-4475-2. Epub 2017 Aug 22. PMID 28831674
- [Background] Chan BK, Wiseberg-Firtell JA, Jois RH, Jensen K, Audisio RA. Localization techniques for guided surgical excision of non-palpable breast lesions. Cochrane Database Syst Rev. 2015 Dec 31;2015(12):CD009206. doi: 10.1002/14651858.CD009206.pub2. PMID 26718728
- [Background] Hu X, Li S, Jiang Y, Wei W, Ji Y, Li Q, Jiang Z. Intraoperative ultrasound-guided lumpectomy versus wire-guided excision for nonpalpable breast cancer. J Int Med Res. 2020 Jan;48(1):300060519896707. doi: 10.1177/0300060519896707. PMID 31937169
- [Background] Ramos M, Diaz JC, Ramos T, Ruano R, Aparicio M, Sancho M, Gonzalez-Orus JM. Ultrasound-guided excision combined with intraoperative assessment of gross macroscopic margins decreases the rate of reoperations for non-palpable invasive breast cancer. Breast. 2013 Aug;22(4):520-4. doi: 10.1016/j.breast.2012.10.006. Epub 2012 Oct 27. PMID 23110817
- [Background] Ahmed M, Douek M. Intra-operative ultrasound versus wire-guided localization in the surgical management of non-palpable breast cancers: systematic review and meta-analysis. Breast Cancer Res Treat. 2013 Aug;140(3):435-46. doi: 10.1007/s10549-013-2639-2. Epub 2013 Jul 23. PMID 23877340
- [Background] Krekel NM, Haloua MH, Lopes Cardozo AM, de Wit RH, Bosch AM, de Widt-Levert LM, Muller S, van der Veen H, Bergers E, de Lange de Klerk ES, Meijer S, van den Tol MP. Intraoperative ultrasound guidance for palpable breast cancer excision (COBALT trial): a multicentre, randomised controlled trial. Lancet Oncol. 2013 Jan;14(1):48-54. doi: 10.1016/S1470-2045(12)70527-2. Epub 2012 Dec 4. PMID 23218662
- [Background] Dogan BE, Whitman GJ. Intraoperative breast ultrasound. Semin Roentgenol. 2011 Oct;46(4):280-4. doi: 10.1053/j.ro.2011.02.009. No abstract available. PMID 22035670
- [Background] Dauphine C, Reicher JJ, Reicher MA, Gondusky C, Khalkhali I, Kim M. A prospective clinical study to evaluate the safety and performance of wireless localization of nonpalpable breast lesions using radiofrequency identification technology. AJR Am J Roentgenol. 2015 Jun;204(6):W720-3. doi: 10.2214/AJR.14.13201. PMID 26001262
- [Background] Look Hong N, Wright FC, Semple M, Nicolae AM, Ravi A. Results of a phase I, non-randomized study evaluating a Magnetic Occult Lesion Localization Instrument (MOLLI) for excision of non-palpable breast lesions. Breast Cancer Res Treat. 2020 Feb;179(3):671-676. doi: 10.1007/s10549-019-05499-z. Epub 2019 Nov 21. PMID 31754951
- [Background] Pieszko K, Wichtowski M, Cieciorowski M, Jamont R, Murawa D. Evaluation of the nonradioactive inducible magnetic seed system Magseed for preoperative localization of nonpalpable breast lesions - initial clinical experience. Contemp Oncol (Pozn). 2020;24(1):51-54. doi: 10.5114/wo.2020.93677. Epub 2020 Mar 13. PMID 32514238
- [Background] Patel SN, Mango VL, Jadeja P, Friedlander L, Desperito E, Wynn R, Feldman S, Ha R. Reflector-guided breast tumor localization versus wire localization for lumpectomies: A comparison of surgical outcomes. Clin Imaging. 2018 Jan-Feb;47:14-17. doi: 10.1016/j.clinimag.2017.07.020. Epub 2017 Aug 1. PMID 28818762
- [Background] Srour MK, Kim S, Amersi F, Giuliano AE, Chung A. Comparison of Multiple Wire, Radioactive Seed, and Savi Scout(R) Radar Localizations for Management of Surgical Breast Disease. Ann Surg Oncol. 2021 Apr;28(4):2212-2218. doi: 10.1245/s10434-020-09159-1. Epub 2020 Sep 28. PMID 32989660
- [Background] Lovrics PJ, Goldsmith CH, Hodgson N, McCready D, Gohla G, Boylan C, Cornacchi S, Reedijk M. A multicentered, randomized, controlled trial comparing radioguided seed localization to standard wire localization for nonpalpable, invasive and in situ breast carcinomas. Ann Surg Oncol. 2011 Nov;18(12):3407-14. doi: 10.1245/s10434-011-1699-y. Epub 2011 Apr 30. PMID 21533657
- [Background] Gray RJ, Salud C, Nguyen K, Dauway E, Friedland J, Berman C, Peltz E, Whitehead G, Cox CE. Randomized prospective evaluation of a novel technique for biopsy or lumpectomy of nonpalpable breast lesions: radioactive seed versus wire localization. Ann Surg Oncol. 2001 Oct;8(9):711-5. doi: 10.1007/s10434-001-0711-3. PMID 11597011
- [Background] McCahill LE, Single RM, Aiello Bowles EJ, Feigelson HS, James TA, Barney T, Engel JM, Onitilo AA. Variability in reexcision following breast conservation surgery. JAMA. 2012 Feb 1;307(5):467-75. doi: 10.1001/jama.2012.43. PMID 22298678
- [Background] Abel TN, Bourke AG. Can micro-computed tomography imaging improve interpretation of macroscopic margin assessment of specimen radiography in excised breast specimens? J Cancer Res Ther. 2020 Oct-Dec;16(6):1366-1370. doi: 10.4103/jcrt.JCRT_949_19. PMID 33342798
- [Background] Spinelle L, Gerboles M, Kok G, Persijn S, Sauerwald T. Review of Portable and Low-Cost Sensors for the Ambient Air Monitoring of Benzene and Other Volatile Organic Compounds. Sensors (Basel). 2017 Jun 28;17(7):1520. doi: 10.3390/s17071520. PMID 28657595
- [Background] Kato S, Post GC, Bierbaum VM, Koch TH. Chemical ionization mass spectrometric determination of acrolein in human breast cancer cells. Anal Biochem. 2002 Jun 15;305(2):251-9. doi: 10.1006/abio.2002.5682. PMID 12054454
- [Background] Kato S, Burke PJ, Koch TH, Bierbaum VM. Formaldehyde in human cancer cells: detection by preconcentration-chemical ionization mass spectrometry. Anal Chem. 2001 Jul 1;73(13):2992-7. doi: 10.1021/ac001498q. PMID 11467545
- [Background] He J, Sinues PM, Hollmen M, Li X, Detmar M, Zenobi R. Fingerprinting breast cancer vs. normal mammary cells by mass spectrometric analysis of volatiles. Sci Rep. 2014 Jun 6;4:5196. doi: 10.1038/srep05196. PMID 24903350
- [Background] Silva CL, Perestrelo R, Silva P, Tomas H, Camara JS. Volatile metabolomic signature of human breast cancer cell lines. Sci Rep. 2017 Mar 3;7:43969. doi: 10.1038/srep43969. PMID 28256598
- [Background] Gouzerh F, Bessiere JM, Ujvari B, Thomas F, Dujon AM, Dormont L. Odors and cancer: Current status and future directions. Biochim Biophys Acta Rev Cancer. 2022 Jan;1877(1):188644. doi: 10.1016/j.bbcan.2021.188644. Epub 2021 Nov 1. PMID 34737023
- [Background] St John ER, Balog J, McKenzie JS, Rossi M, Covington A, Muirhead L, Bodai Z, Rosini F, Speller AVM, Shousha S, Ramakrishnan R, Darzi A, Takats Z, Leff DR. Rapid evaporative ionisation mass spectrometry of electrosurgical vapours for the identification of breast pathology: towards an intelligent knife for breast cancer surgery. Breast Cancer Res. 2017 May 23;19(1):59. doi: 10.1186/s13058-017-0845-2. PMID 28535818
- [Background] Pleijhuis RG, Graafland M, de Vries J, Bart J, de Jong JS, van Dam GM. Obtaining adequate surgical margins in breast-conserving therapy for patients with early-stage breast cancer: current modalities and future directions. Ann Surg Oncol. 2009 Oct;16(10):2717-30. doi: 10.1245/s10434-009-0609-z. Epub 2009 Jul 17. PMID 19609829
- [Background] Ranganathan K, Singh P, Raghavendran K, Wilkins EG, Hamill JB, Aliu O, Newman LA, Hutton D, Momoh AO. The Global Macroeconomic Burden of Breast Cancer: Implications for Oncologic Surgery. Ann Surg. 2021 Dec 1;274(6):1067-1072. doi: 10.1097/SLA.0000000000003662. PMID 32097168
- [Background] Cid C, Herrera C, Rodriguez R, Bastias G, Jimenez J. [Assessing the economic impact of cancer in Chile: a direct and indirect cost measurement based on 2009 registries]. Medwave. 2016 Aug 2;16(7):e6509. doi: 10.5867/medwave.2016.07.6509. Spanish. PMID 27532152
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer Statistics, 2021. CA Cancer J Clin. 2021 Jan;71(1):7-33. doi: 10.3322/caac.21654. Epub 2021 Jan 12. PMID 33433946
- [Background] Piper ML, Wong J, Fahrner-Scott K, Ewing C, Alvarado M, Esserman LJ, Mukhtar RA. Success rates of re-excision after positive margins for invasive lobular carcinoma of the breast. NPJ Breast Cancer. 2019 Sep 6;5:29. doi: 10.1038/s41523-019-0125-7. eCollection 2019. PMID 31508489